CLINICAL TRIAL: NCT06850181
Title: "The Effect of Game-Based Practices on the Gaming Experience and Learning Motivation of Students in Psychiatric Nursing Courses"
Brief Title: Gaming Experience and Learning Motivation of Students in Psychiatric Nursing Courses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tuba Çömez İkican, Asisstan Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/565
Record Dates: First submitted 2025-02-06; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Game-Based Learning; Nursing Students; Nursing Education; Motivation
Keywords: Game-based learning, Nursing education, Learning motivation, Gaming experience, Undergraudate nursing student;

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Behavioral: game experience and learning motivation

INTERVENTIONS:
Behavioral: game experience and learning motivation — game experience and learning motivation

SUMMARY:
This research is carried out by Dr Tuba Çömez İkican, Dr. Olga İncesu, Dr. Gizem Şahin Bayındır. In this research aimed to determine the effect of game-based applications in nursing education on students' game experience and learning motivation.

H1: 'Game-based practices significantly increase the game experiences of students taking psychiatric nursing course.' H2: 'Game-based practices significantly increase the learning motivation of students taking psychiatric nursing course.' The population of the study consisted of all 3rd year students (N=69) studying in a nursing faculty in Istanbul in the 2024-2025 academic year and taking the Mental Health and Diseases Nursing course. After the purpose of the study was explained, 68 students who gave written and verbal consent to participate in the study were included in the sample.

The research is a quasi-experimental research design with pre-test / post-test control.

Inclusion Criteria

* To be enrolled in Mental Health and Diseases Nursing course
* Not working as a part/full-time nurse
* To be 18 years of age or older,
* To agree to participate in the research,
* Continuing to attend lectures and laboratory applications

Data will be collected through the Personel Information Form, Gameful Experience Scale, Motivated Strategies for Learning Questionnaire. The personel information form was prepared by the researchers in line with the literature. Permission was obtained from the scale owners for the scales to be used in the study.

Institutional permission from Istanbul University School of Nusing and ethics committee approval (Number: 14.11.2024-1142952) from Istanbul University- Cerrahpasa Social and Human Sciences Research Ethics Committee obtained in order to conduct the study. Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 29). The expenses of the research will be covered by the researcher.

DETAILED DESCRIPTION:
In recent years, the gaming experience has become an effective practice that contributes to individuals' cognitive and emotional development beyond mere entertainment. Game-based applications aim to enhance students' motivation, willingness to learn, and achievement levels while making education more engaging and enjoyable. Nursing students need to produce rapid and effective solutions when interacting with patients or making clinical decisions. Gaming experiences, particularly those focused on strategy and problem-solving themes, can improve such thinking skills and boost their motivation. Although studies using gamification methods in nursing education exist, no study has been found that evaluates game-based learning experiences or explores the relationship between game-based learning and willingness to learn. This research aims to determine the impact of game-based applications in nursing education on students' gaming experiences and their learning motivation.

In this research aimed to determine the effect of game-based applications in nursing education on students' game experience and learning motivation.

H1: 'Game-based practices significantly increase the game experiences of students taking psychiatric nursing course.' H2: 'Game-based practices significantly increase the learning motivation of students taking psychiatric nursing course.' The population of the study consisted of all 3rd year students (N=69) studying in a nursing faculty in Istanbul in the 2024-2025 academic year and taking the Mental Health and Diseases Nursing course. After the purpose of the study was explained, 68 students who gave written and verbal consent to participate in the study were included in the sample.

Dependent Variables: Game Playing Experience Scale score, Motivation and Learning Strategies Scale score Independent Variables: Sociodemographic characteristics of the participants

The research is a quasi-experimental research design with pre-test / post-test control.

Inclusion Criteria

* To be enrolled in Mental Health and Diseases Nursing course
* Not working as a part/full-time nurse
* To be 18 years of age or older,
* To agree to participate in the research,
* Continuing to attend lectures and laboratory applications

The study was conducted at Istanbul University Faculty of Nursing between November 2024 and December 2024.Data will be collected through the Personel Information Form, Gameful Experience Scale, Motivated Strategies for Learning Questionnaire. The personel information form was prepared by the researchers in line with the literature. Permission was obtained from the scale owners for the scales to be used in the study.

* Socio-Demographic Characteristics Form: This form consists of a total of 8 questions including sociodemographic characteristics developed by the researchers within the framework of the literature.
* Game Playing Experience Scale: The scale was developed by Eppman et al. in 2018 and Çömez et al. in 2024. Turkish validity and reliability was conducted by İkican et al. The scale, which aims to measure the participants' experiences about the game, consists of a total of 27 items and 5 sub-dimensions. A 5-point Likert scale is used in the evaluation of the scale. Items 18, 21, 22 and 23 in the scale are scored inversely ('Never' - 5, 'Rarely' - 4, 'Occasionally' - 3, 'Often' - 2 and 'Always' - 1). The internal consistency coefficient (cronbach alpha) of the scale was found to be 0.89.
* Motivation and Learning Strategies Scale: The scale was developed by Pintrich, Smith, Garcia, and McKeachie (1991) to measure 'the different learning strategies and motivational orientations that university students use towards a university course based on their self-reports'. The Turkish validity and reliability of the scale was conducted by Büyüköztürk, Akgün, Kahveci and Demirel in 2004. The scale consists of two parts: learning strategies scale and motivation scale. consists of the Motivation Scale. The part that will be used in this study is the Motivation Scale. The scale consists of internal goal organisation (4 items), external goal organisation (4 items), task value (6 items), self-efficacy related to learning and performance (8 items), self-efficacy related to learning control belief (4 items), test anxiety (5 items), and a total of 6 factors and 31 items. The scale is a 7-point Likert scale ranging from 'absolutely wrong for me (1)' to 'absolutely right for me (7)'.

In the study, the data collection process began after obtaining ethics committee approval and institutional permission. Nursing students who meet the inclusion criteria will be identified, and data will be collected twice as pre-test and post-test. The data collection process is as follows:

Pre-Gaming Experience: Before the intervention, the Socio-Demographic Characteristics Form, Gaming Experience Scale, and Motivation and Learning Strategies Scale will be administered as a pre-test to all students who provide written and verbal consent and meet the inclusion criteria.

Intervention: Over a total of 6 weeks, at the end of each mental health and psychiatric nursing class, questions related to the week's topic will be presented using an online assessment and evaluation tool (quiz program) with visual aids. During the first week of the lab program, a role-play exercise and its features will be explained, and a demonstration video will be shown to the students. For the following 5 weeks, students will be asked to perform group role-play activities based on assigned case scenarios.

Post-Intervention: At the end of the 6th week, the Gaming Experience Scale and Motivation and Learning Strategies Scale will be re-administered to the students as a post-test.

Institutional permission from Istanbul University School of Nusing and ethics committee approval (Number: 14.11.2024-1142952) from Istanbul University- Cerrahpasa Social and Human Sciences Research Ethics Committee obtained in order to conduct the study. Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 29). The expenses of the research will be covered by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in Mental Health and Diseases Nursing course
* Not working as a part/full-time nurse
* To be 18 years of age or older,
* To agree to participate in the research,
* Continuing to attend lectures and laboratory applications

Exclusion Criteria:

* Be less than 18 years old,

  * Not knowing how to read, write and speak Turkish,
  * Having any cognitive, sensory and spiritual problems,
  * Not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Socio-Demographic Characteristics Form | Baseline
  Socio-Demographic Characteristics Form: This form consists of a total of 8 questions including sociodemographic characteristics developed by the researchers within the framework of the literature.
Game Playing Experience Scale | Baseline
  Game Playing Experience Scale: The scale, which aims to measure the participants' experiences about the game, consists of a total of 27 items and 5 sub-dimensions.
Motivation and Learning Strategies Scale | Baseline
  Motivation and Learning Strategies Scale: The scale was developed to measure 'the different learning strategies and motivational orientations that university students use towards a university course based on their self-reports'.

SECONDARY OUTCOMES:
Game Playing Experience Scale | 6 weeks
  Game Playing Experience Scale. The scale, which aims to measure the participants' experiences about the game, consists of a total of 27 items and 5 sub-dimensions.
Motivation and Learning Strategies Scale | 6 weeks
  Motivation and Learning Strategies Scale: The scale was developed to measure 'the different learning strategies and motivational orientations that university students use towards a university course based on their self-reports'.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 5- Blanco, A, Torente, J, Manjon, FB, Ruiz, P, Giner M. (2017). "Using A Videogame To Facilitate Nursing And Medical Students' First Visit To The Operating Theatre. A Randomized Controlled Trial". Nurse Educ Today, (55), 45-53. 6- Garrison, E., Colin, S., Lemberger, O., & Lugod, M. (2021). Interactive learning for nurses through gamification. JONA: The Journal of Nursing Administration, 51(2), 95-100.
- [Result] 1- Garrison, E., Colin, S., Lemberger, O., & Lugod, M. (2021). Interactive learning for nurses through gamification. JONA: The Journal of Nursing Administration, 51(2), 95-100. 2- Lee, M. D. (2016). Gamification and the psychology of game design in transforming mental health care. Journal of the American Psychiatric Nurses Association, 22(2), 134-136. 3- Zugai, J. S., Orr, F., & Levett-Jones, T. (2021). Online Gamified Quizzes in Undergraduate Mental Health Nursing Education: Thematic Analysis of Students' Qualitative Views. Issues in Mental Health Nursing, 1-5. 4- Zichermann, G. ve Cunningham, C. (2011). Gamification by design: Implementing game mechanics in web and mobile apps. O'Reilly Media, Inc.